CLINICAL TRIAL: NCT01062854
Title: Effects of Earplugs on Sleep and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ronald D. Chervin, M.D., M.S., Michael S Aldrich Collegiate Professor of Sleep Medicine and Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HUM00023548
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Sleep Disordered Breathing
Keywords: snoring, sleep disordered breathing, polysomnography, sleep fragmentation
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Earplugs (Experimental): Subjects randomized to this arm of the study will wear earplugs during their baseline sleep study (polysomnogram).
  Interventions: Other: Soft earplugs are worn during sleep study
- Comparison group (No Intervention): Subjects randomized to the comparison arm will not wear earplugs during their baseline sleep study.

INTERVENTIONS:
Other: Soft earplugs are worn during sleep study — Subjects are asked to wear earplugs when possible for 3-5 nights prior to their baseline sleep study. On the night of their sleep study they are randomized to either "wears earplugs" or "no earplugs" groups.
  Other Names: Howard Leight (Sperian) Max-1/3303361 uncorded earplugs, NRR33, SNR 37dB
  Arms: Earplugs

SUMMARY:
The main goal of this study is to assess whether use of earplugs has any effect on sleep, sleep apnea, and daytime sleepiness in individuals who snore.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18 or older
* Scheduled at the University of Michigan Sleep Disorders Center for a diagnostic polysomnogram to evaluate for sleep-disordered breathing

Exclusion Criteria:

* Medical, psychiatric or other conditions that would interfere with interpretation of the results of the sleep studies or the subject's ability to complete the Stanford Sleepiness Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sleep measures (rates of apneas and hypopneas, oxygen desaturation, arousals, sleep stages, respiratory cycle-related EEG changes [RCREC]) | up to 2 years after the sleep study

SECONDARY OUTCOMES:
Subjective sleepiness measures (Stanford Sleepiness Scale) | on awakening after the sleep study

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Sleep Disorders Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Chirakalwasan N, Ruzicka DL, Burns JW, Chervin RD. Do snoring sounds arouse the snorer? Sleep. 2013 Apr 1;36(4):565-71. doi: 10.5665/sleep.2546. PMID 23565002